CLINICAL TRIAL: NCT00970073
Title: A Randomized Controlled Clinical Trial of Low Dose Thymoglobulin and Extended Delay of Calcineurin Inhibitor Therapy for Renal Protection After Liver Transplantation
Brief Title: Low Dose Thymoglobulin to Protect Kidney Function After Liver Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Bijan Eghtesad, MD, HPBT Staff Surgeon, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCIRB 09-432
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Liver Transplantation
Keywords: calcineurin inhibitor delay; Kidney
MeSH Terms: interventions — thymoglobulin; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Delayed CNI Group 1 (Experimental): Thymoglobulin 3mg total, administered on Days 0 and 2 (after transplant), plus MMF and corticosteroids. CNI administration delayed until 10 days post transplant. tacrolimus 3-8 (trough concentration)
  Interventions: Biological: Thymoglobulin 3mg total; Drug: Mycophenolate mofetil; Drug: tacrolimus 3-8
- Delayed CNI Group 2 (Experimental): Thymoglobulin 4.5mg total, plus MMF and corticosteroids. CNI therapy delayed until 10 days post transplant.tacrolimus 3-8 (trough concentration)
  Interventions: Biological: Thymoglobulin 4.5mg total; Drug: Mycophenolate mofetil; Drug: tacrolimus 3-8
- Early CNI / Control Arm (Active Comparator): Standard post liver transplant therapy to include: tacrolimus 8-12 (trough concentration) initiated within 48 hours post-transplant, plus mycophenolate mofetil (MMF) and corticosteroids to be administered within 24 hours after transplant (Day 0).
  Interventions: Drug: Mycophenolate mofetil; Drug: tacrolimus 8-12

INTERVENTIONS:
Biological: Thymoglobulin 3mg total — 1.5 mg/kg induction on Day 0 and 1.5 mg/kg induction on Day 2 (total of 3 mg/kg)
  Arms: Delayed CNI Group 1
Biological: Thymoglobulin 4.5mg total — 1.5 mg/kg induction on Days 0, 2 and 4 (total 4.5 mg/kg)
  Arms: Delayed CNI Group 2
Drug: Mycophenolate mofetil — 1000 mg PO/IV BID for up to 6 months
  Other Names: CellCept
Drug: tacrolimus 3-8 — Trough concentration between 3 ng/mL and 8 ng/mL starting on Day 10 and continuing beyond Day 180
  Other Names: Prograf
  Arms: Delayed CNI Group 1; Delayed CNI Group 2
Drug: tacrolimus 8-12 — Trough concentration between 8 ng/mL and 12 ng/mL on Days 0-10; between 6 ng/mL and 12 ng/mL on Days 10-30; between 6 ng/mL and 10 ng/mL Days 31-60; between 5 ng/mL and 8 ng/mL Days 61-179; and between 3 ng/mL and 8 ng/mL beyond Day 180.
  Other Names: Prograf
  Arms: Early CNI / Control Arm

SUMMARY:
This study will evaluate the use of a drug called Thymoglobulin, combined with a delayed start of the anti-rejection drugs (10 days after liver transplant), compared to the current approach of starting anti-rejection drugs called calcineurin inhibitors or CNI's within 2 days after the liver transplant.

DETAILED DESCRIPTION:
Strong anti-rejection drugs like tacrolimus or cyclosporine, are given to patients who have received transplants, to ensure that the patient's body does not reject the new organ. In some cases, while anti-rejection medications protect a newly transplanted liver, they can injure the patient's kidneys and cause them not to work as well as they should. The purpose of this pilot study is to determine the best way to protect kidney function and to ensure that the newly transplanted liver is not rejected. This study will evaluate the use of a drug called Thymoglobulin, combined with a delayed start of the anti-rejection drugs (10 days after liver transplant), compared to the current approach of starting anti-rejection drugs called calcineurin inhibitors or CNI's within 2 days after the liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing deceased donor solitary liver transplantation
* Adults aged 18-70 at time of transplantation
* Hepatocellular carcinoma as indication for OLT within the Milan Criteria
* Hepatitis C positive or negative patients
* Willingness to comply with study procedures
* Able to sign informed consent

Exclusion Criteria:

* Prior kidney transplantation
* Congenital or iatrogenic absence of one kidney
* Subjects on renal replacement therapy at the time of OLT
* MELD score > 28
* HIV positive patient
* Patient with current severe systemic infection
* History of bacterial peritonitis within 30 days prior to OLT
* Active infection or recent infection within 30 days prior to OLT
* Use of calcineurin inhibitor continuously for more than 90 days within the past 6 months
* History of hypersensitivity to thymoglobulin, rabbits, tacrolimus or iohexol
* Women of childbearing age who are unwilling to use effective contraceptive methods during the duration of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Eghtesad, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic (Main Campus), Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Delayed CNI Group 1 | Delayed CNI Group 2 | Early CNI / Control Arm
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed CNI Group 1 | Delayed CNI Group 2 | Early CNI / Control Arm | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 10 | 28
  >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 6
  Male | 8 | 9 | 7 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Estimated Glomerular Filtration Rate (eGFR) at 12 Months Post-surgery
Description: Postoperative acute kidney injury is measured as reduced (eGFR) within 12 months post-surgery.
Time Frame: 12 Months
Measure: Median (90% Confidence Interval); unit: mL/min
Arm/Group | Delayed CNI Group 1 | Delayed CNI Group 2 | Early CNI / Control Arm
Number analyzed (Participants) | 10 | 10 | 10
mL/min | 72 [57.7 to 86.3] | 87.8 [67.3 to 108.3] | 51.0 [24.4 to 77.6]

2. Secondary Outcome: Patient Survival
Time Frame: 12 months post-transplant
Population: Kaplan- Meier
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed CNI Group 1 | Delayed CNI Group 2 | Early CNI / Control Arm
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 9 | 8

3. Secondary Outcome: Graft Survival
Description: 90% graft survival, related to the deaths of 3 patients during the study period.
Time Frame: 12 months post transplant
Population: Kaplan Meier for patient survival
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed CNI Group 1 | Delayed CNI Group 2 | Early CNI / Control Arm
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 9 | 8

4. Secondary Outcome: Allograft Rejection Rates at 30 Days
Description: Acute Allograft Rejection
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed CNI Group 1 | Delayed CNI Group 2 | Early CNI / Control Arm
Number analyzed (Participants) | 10 | 10 | 10
Participants | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Delayed CNI Group 1 | Delayed CNI Group 2 | Early CNI / Control Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/10 | 2/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 2/10 | 5/10 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed CNI Group 1 (N=10) | Delayed CNI Group 2 (N=10) | Early CNI / Control Arm (N=10)
Metastatic Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Graft vs Host Disease (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed CNI Group 1 (N=10) | Delayed CNI Group 2 (N=10) | Early CNI / Control Arm (N=10)
HCV recurrence (Infections and infestations) | 2 (2) | 5 (5) | 4 (4) — HCV recurrence in HCV positive recipients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes